CLINICAL TRIAL: NCT01800474
Title: A Non-interventional Study to Evaluate the Use of Pliaglis in Daily Practice
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: 05PT1209
Record Dates: First submitted 2013-01-18; First posted 2013-02-27 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2015-02

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
A multe-center, non-interventional study in Europe to evaluate Pliaglis in daily practice

DETAILED DESCRIPTION:
A multi-center, non-interventional study, including up to 700 subjects at approximately 70 sites in 5 European countries to evaluate the post-market safety profile of Pliaglis and the efficacy of Pliaglis in terms of pain reduction, satisfaction with the product and daily practice use prior to pre-defined aesthetic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient treated with Pliaglis by the Investigator or other healthcare professional according to label (refer to SmPC)
* Patient had already consented to receive any one or more of the following aesthetic procedures after Pliaglis administration:

  1. Pulsed-dye laser therapy
  2. Laser-assisted hair removal
  3. Non-ablative laser resurfacing
  4. Dermal filler injection
  5. Vascular access

Exclusion Criteria:

* Patient treated with other injectable or topical anaesthetic(s) for the pre-defined aesthetic procedure
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient aiming to perform one or more of the following aesthetic procedures:
  1. Pulsed-dye laser therapy
  2. Laser-assisted hair removal
  3. Non-ablative laser resurfacing
  4. Dermal filler injection
  5. Vascular access
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Post-market safety profile of Pliaglis assessed on spontaneously reported Adverse Reactions | After Pliaglis application and throughout the site visit (day of application)

SECONDARY OUTCOMES:
Efficacy of Pliaglis | After completing Pliaglis treatment and procedure, i.e. at the end of the site visit (day of application)
  Pain intensity by VAS, satisfaction with pain reduction, willingness to re-use/recommend Pliaglis

CONTACTS AND LOCATIONS:
Overall Officials: Max Murison, Dr., Principal Investigator — National coordinating investigator; Maurizio Podda, Dr, Principal Investigator — National coordinating investigator; Hugues Cartier, Dr, Principal Investigator — National coordinating investigator; Carlos Guillén, Dr, Principal Investigator — National coordinating investigator
Locations (4):
- Centre Médical Saint-Jean, Arras, France
- Klinikum Darmstadt Hautklinik, Darmstadt, Germany
- Clínica Dermatológica Dr. Guillén, Valencia, Spain
- Swansea Laser Clinic, Swansea, United Kingdom

REFERENCES:
- [Derived] Jain R, Arias GM, Naranjo P, Murison M, Lopez Estebaranz JL, Fratila A, Prager W, Barona CG, Weidmann M, Dahan S, Cartier H, Sattler G, Podda M. The Use of a Self-Occluding Topical Anasthetic in Daily Practice: A Non-Interventional Study. J Drugs Dermatol. 2018 Apr 1;17(4):413-418. PMID 29601618